CLINICAL TRIAL: NCT05242588
Title: A Randomized, Double-blind, Placebo-controlled, Phase II, Multicenter Study to Evaluate the Preliminary Efficacy, Safety, and Pharmacokinetics of Subcutaneous JS005 in Chinese Adults With Active Non-radiographic Axial Spondyloarthritis
Brief Title: Evaluate the Preliminary Efficacy, Safety, and PK of Subcutaneous JS005 in Chinese Adult Patients With Active Nr-axSpA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS005-004-II-nr-axSpA
Record Dates: First submitted 2021-11-30; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Non-radiographic Axial Spondyloarthritis
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator
Masking Description: Priticipant,Care provider and investigators are masked in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- JS005 150 mg (Experimental): 30 patients will be enrolled in this arm.
  Interventions: Biological: JS005
- Placebo 150 mg (Placebo Comparator): 10 patients will be enrolled in this arm.
  Interventions: Biological: Placebo
- JS005 300 mg (Experimental): 30 patients will be enrolled in this arm.
  Interventions: Biological: JS005
- Placebo 300 mg (Placebo Comparator): 10 patients will be enrolled in this arm.
  Interventions: Biological: Placebo
- JS005 450 mg (Experimental): 30 patients will be enrolled in this arm.
  Interventions: Biological: JS005
- Placebo 450 (Placebo Comparator): 10 patients will be enrolled in this arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: JS005 — 30 subjectes in JS005 150mg chort, JS005 300mg chort, and JS005 450mg chort receive JS005 150mg, JS005 300mg and JS005 450mg subcutaneous injection seperately at Week 0, 1, 2, and 3, and monthly dose starting at Week 4 (dosing in Week 4, 8, and 12).
  Other Names: Recombinant humanized anti-IL-17A monoclonal antibody injection
  Arms: JS005 150 mg; JS005 300 mg; JS005 450 mg
Biological: Placebo — 10 subjects in JS005 150mg chort, JS005 300mg chort, and JS005 450mgchort receive the placebo subcutaneous injection seperately at Week 0, 1, 2, and 3, and monthly dose starting at Week 4 (dosing in Week 4, 8, and 12).
  Arms: Placebo 150 mg; Placebo 300 mg; Placebo 450

SUMMARY:
The purpose of this study is to evaluate preliminary efficacy, safety pharmacokinetic (PK) characteristics, pharmacodynamics (PD) haracteristics and immunogenicity of JS005 at different doses in Chinese patients with active non-radiographic axial spondyloarthritis(nr-axSpA). Treatment difference of JS005 150mg,300mg,450mg vs. placebo in Chinese nr-axSpA patients in terms of ASAS 40 response rate at Week 16 as well as safety profile will be provided by the study .

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study. Approximately 120 patients who meet the eligibility criteria will be randomized to one of three treatment cohorts (JS005 150 mg, 300 mg, 450mg in a ratio of 1:1:1),then using secondary randomization method, 40 patients in each group will be randomized in a 3: 1 ratio to receive investigational product or placebo.

1. JS005 150mg Cohort: JS005 150 mg or placebo treatment(JS005:Placrbo=3:1) s.c. prefilled syringe (PFS) on Week 0, 1, 2, 3, 4,8 and 12
2. JS005 300mg Cohort: JS005 300 mg or placebo treatment(JS005:Placrbo=3:1) s.c. PFS on Week0, 1, 2 ,3, 4,8,and 12 3 .JS005 450mg Cohort: JS005 450 mg or placebo treatment(JS005:Placrbo=3:1) s.c. PFS on Week0, 1, 2 ,3, 4,8,and 12 Based on the clinical judgment of disease activity by the investigator and the patient, background medications, such as NSAIDs and DMARDs, may have been modified or added to treat signs and symptoms of nr-axSpA from Week 16 on.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who do not meet the modified New York criteria for AS in 1984; Meet the 2009 axSpA classification criteria recommended by International Assessment Society of Axial Spondyloarthritis (ASAS): inflammatory back pain for at least 3 months; Age of onset < 45 years; Sacroiliitis on MRI with≥ 1 axial spondyloarthritis features or HLA-B27 positive with ≥ 2 SpA features (MRI and X-ray of sacroiliac joint as confirmed by central readers).
2. Objective signs of inflammation at screening: active inflammation of the sacroiliac joints on MRI and/or high sensitivity C-reactive protein (hsCRP) > upper limit of normal without other diagnoses to explain the MRI results or elevated hsCRP.
3. Active axSpA at screening and baseline: assessed by total Bath ankylosing spondylitis disease activity index (BASDAI) ≥ 4 (0-10 scale) and spinal pain ≥ 4 (according to the 0-10 NRS scale, BASDAI question #2).
4. Voluntarily participate in this clinical trial and sign the informed consent form.
5. Male or female aged between 18 and 65 years (both inclusive) at the time of signing informed consent. Female subjects of childbearing age are required to have a confirmed negative result of urine and/or serum pregnancy test performed within 3 days before randomization and agree to use reliable contraceptive measures during the study; Male subjects and their female partners of childbearing age must agree to use reliable contraception during the study.
6. Patients meet at least one of the following: 1) have an inadequate or ineffective response to NSAIDs, 2) have been intolerant to at least one dose of NSAIDs, 3) have contraindications to NSAIDs therapy. Inadequate or ineffective response to NSAIDs is defined as no remission after continuous treatment with standard doses of at least 2 NSAIDs for a total of no less than 4 weeks and no less than 2 weeks for each NSAID.
7. Patients regularly taking NSAIDs as part of their AS therapy are required to maintain a stable dose for at least 2 weeks prior to randomization.
8. Patients using tumor necrosis factor α (TNFα) inhibitors must have experienced an inadequate response to the standard treatment dose for at least 3 months, or have been intolerant to TNFα inhibitors.

Exclusion Criteria:

1. Unable or unwilling to undergo MRI.
2. Previous exposure to JS005 or any other biologic drug directly targeting IL-17 or IL-17 receptor.
3. Have taken high potency analgesics (e.g., opiates of methadone, hydromorphone, morphine) within 2 weeks prior to randomization.
4. Previous treatment with any intra-articular injection (e.g., glucocorticoids) within 4 weeks prior to randomization.
5. Previous treatment with any biological immunomodulating agents other than the TNFα inhibitors.
6. Treatment with JAK inhibitor agents within 8 weeks prior to randomization and unwilling to discontinue during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of nr-axSpA patients meeting the Assessment of Spondylo Arthritis international Society (ASAS) 40 response criteria | From week 0 to week 16
  at the end of treatment Week 16 .

SECONDARY OUTCOMES:
ASAS20 response criteria | From week 0 to week 16
  The proportion of patients meeting the ASAS20 response criteria at the end of treatment Week 16
ASAS 5/6 response criteria | From week 0 to week 16
  The proportion of patients meeting the ASAS 5/6 response criteria at the end of treatment Week 16;
High-sensitivity C-reactive protein (hsCRP) | From week 0 to week 16
  The change from baseline in high-sensitivity C-reactive protein (hsCRP) at the end of treatment Week 16
The inflammation score of the sacroiliac joint | From week 0 to week 16
  The change from baseline in the inflammation score of the sacroiliac joint by MRI at the end of treatment Week 16
Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) | From week 0 to week 16
  The change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) at the end of treatment Week 16;
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | From week 0 to week 16
  The change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at the end of treatment Week 16
Bath Ankylosing Spondylitis Functional Index (BASFI) | From week 0 to week 16
  The change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at the end of treatment Week 16
Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) | From week 0 to week 16
  The change from baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at the end of treatment Week 16
Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) | From week 0 to week 16
  The change from baseline in Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) at the end of treatment Week 16
The patient's global assessment of disease activity | From week 0 to week 16
  Numeric Rating Scale (NRS, ranging from 0 not active to 10 very active) will be used to evaluate the patient's global assessment of disease activity. Patient will be asked by one question: How active was your spondylitis on average during the last week？
The patient's assessment of inflammatory back pain intensity | From week 0 to week 16
  NRS(ranging from 0 no pain to 10 most severe pain) will be used to assess the patient's inflammatory back pain intensity. The assessment is based on two questions: "Based on your assessment, please indicate How much pain of your spine due to AS do you have ?" and "Based on your assessment, please specify How much pain of your spine due to AS do you have at night?" When responding, the subject is to consider the average amount of pain in the last week.
ASAS partial remission criteria | From week 0 to week 16
  The proportion of patients meeting ASAS partial remission criteria at the end of treatment Week 16

OTHER OUTCOMES:
Pharmacokinetic endpoint | From Baseline to week 24,Total 24 weeks
  • Population pharmacokinetic analysis of plasma concentrations will be performed to explore the exposure of JS005 in patients and the influencing factors of exposure
Pharmacodynamic endpoint | From Baseline to week 24,Total 24 weeks
  • Concentrations and the changes of free and/or total IL-17 in serum before and after administration.
Immunogenicity endpoint | From Baseline to week 24,Total 24 weeks
  • Anti-drug antibody (ADA), for the ADA positive samples, it is necessary to test the titer and determine whether it is a neutralizing antibody (Nab).
Safety evaluation | From V1 to V12, Total 36 Weeks
  Safety evaluation will be documented as numbers of adverse event(AE).

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen Memorial Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Nanfang Medical University, Guangzhou, Guangdong
  - Shantou University Medical Collge No.1 Affiliated Hospital, Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Pking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital,Tongji Medical College of HUST, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affilated Hospital of Inner Mongdlia Medical University, Hohhot, Inner Mongolia
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - North Sichuan Medical College Affiliated Hospital, Nanchong, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University,School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
Undecided